CLINICAL TRIAL: NCT07122557
Title: Real World Effectiveness of Bictegravir/Emtricitabine/Tenofovir Alafenamide(BIC/FTC/TAF) in PLWH in Precarity Settings in France
Brief Title: Real World Effectiveness of Bictegravir/Emtricitabine/Tenofovir Alafenamide(BIC/FTC/TAF) in PLWH in Precarity Settings in France -IMEA073
Acronym: PRECARITY
Status: Not yet recruiting | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Other Study IDs: IMEA
Record Dates: First submitted 2025-04-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HIV-1; Public Universal Healthcare Insurance Coverage; BIC/FTC/TAF; Low Income Population
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment naive,virologically suppressed and unsuppressed treatment experienced in 2nd line
  Interventions: Drug: Biktarvy

INTERVENTIONS:
Drug: Biktarvy — this study applies secondary use of data collected from medical health records

SUMMARY:
In France, French citizens with an annual income less than 10339 euros are considered living with low-income and are eligible to benefit from a public universal healthcare insurance coverage called C2S (complémentaire santé solidaire). C2S covers primary care and hospital care. Non-citizens with low income, like some migrants, can also benefit from a public healthcare insurance coverage called AME ("Aide Medicale d'Etat" for State Medical Aid). These criteria are used as a marker of precarity settings (i.e., socio-economic vulnerability) in France. In France, HIV-related care and treatments are reimbursed at 100% (ALD30), whatever the level of precariousness. ART adherence has been shown significantly lower in PLWH with C2S health insurance coverage. Although BIC/FTC/TAF is a recommended preferred option in naive PLWH and in switch or maintenance therapy in most settings, due to the forgiveness profile and the high genetic barrier to resistance, boosted darunavir (DRV/r) remains even more widely used than 2nd generation InSTIs in populations in precarity settings, and Real World Effectiveness (RWE) with BIC/FTC/TAF is missing to better support its use in these settings.

Paris Bichat Hospital (located in one of the poorest districts in the Ile-de-France region) and Nantes university hospital (West France region) follow a cohort of PLWH with a high proportion of populations in precarity settings (i.e with C2S and AME health insurance coverage): Paris Bichat hospital: N=5143 PLWH (December 2021), sex ratio F/M 37/56%, Transgender Women 7%, and born in sub-Saharan African countries 49%. Nantes university hospital: N=2227 PLWH (December 2021), sex ratio F/M 35/65% and born in sub-Saharan African countries 33%. In this cohort of 7370 PLWH in both sites 50% are receiving an InSTI-based ART regimen, regardless of prior treatment history, and at least 40% are receiving care through the C2S or AME, respectively.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients > 18 years during the observation period
* PLWH with C2S or AME heath insurance coverage information available during the observation period
* Treatment naive (TN) on BIC/FTC/TAF OR Treatment experienced virologically suppressed (VS TE) or virologically unsupressed (VU TE) in 2d line BIC/FTC/TAF
* Had at least one follow-up visit after baseline

Exclusion Criteria:

* Missing information regarding health insurance coverage
* On regimen other than BIC/FTC/TAF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naïve (TN) and Virologically Suppressed Treatment Experienced (VS TE) in 2d line treatment, or Virologically Unsuppressed Treatment Experienced (VU TE) in 2d line treatment patients within Paris Bichat and CHU Nantes hospitals who were covered by C2S/AME heath insurance during study period.
  - Those using BIC/FTC/TAF We will conduct descriptive analyses only. Analyses will be disaggregated by TN, VS TE, and VU TE groups.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
i. HIV RNA ≥50 copies/mL at week 48 within the time window OR One HIV RNA ≥50 copies/mL followed by treatment discontinuation before week 48 after reaching HIV RNA < 50 copies/mL | Week 48
ii. Discontinuation due to treatment related adverse event | week 48
iii. Discontinuation due to non-treatment related adverse event, death or other reasons | week 48
iv. On study but missing data in window | Week 48+/- 8 weeks
i. Two consecutive HIV RNA VL ≥200 copies/mL after reaching a HIV RNA < 50 copies/mL | week 48
ii. One HIV RNA VL ≥200 copies/mL followed by baseline treatment discontinuation after reaching HIV RNA < 50 copies/mL | week 48
iii. HIV RNA VL ≥200 copies/mL at week 48 and no other value for confirmation | week 48

SECONDARY OUTCOMES:
• Evaluate the time to treatment discontinuation and reason for discontinuation with BIC/FTC/TAF among TN, VS TE and VU TE PLWH. | week 48
• Describe subsequent regimens among individuals discontinued BIC/FTC/TAF among TN, VS TE and VU TE. | week 48
• Describe the number of hospital medical HIV appointments, and participants baseline characteristics with BIC/FTC/TAF among TN, VS TE and VU TE PLWH | week 48
• Describe treatment emergent resistance profile among participants with confirmed virologic failure with BIC/FTC/TAF among TN, VS TE and VU TE PLWH. | week 48
• Describe the change of CD4 | week 48
  CD4 description
• Factors associated with virologic suppression (HIV RNA<50 copies/mL, FDA Snapshot), confirmed virologic failure (HIV RNA ≥200 copies/mL), discontinuation, and emergence of resistance-associated mutations at failure among TN, VS TE and VU TE. | week 48
• Describe the change of CD8 cell counts | Week 48
  CD8 description
• Describe the change CD4/CD8 ratio | Week 48
  description CD4/CD8 ratio
• Describe the change of BMI | Week 48
  BMI description
• Describe the change of body weight | Week 48
  Body weight description

CONTACTS AND LOCATIONS:
Overall Officials: Roland LANDMAN, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP